CLINICAL TRIAL: NCT00724451
Title: Prospective, Observational, Multicentre Study Evaluating HCV Patients Characteristics of Eligibility and Disease Management in Real Clinical Practice
Brief Title: Observational Study Assessing Chronic Hepatitis C Management in Clinical Practice in Italy (Study P05488 AM1)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05488
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C; Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Chronic Hepatitis C (CHC): Peginterferon-naïve participants with CHC seen in general clinical practice in Italy and treated with either pegylated interferon alfa-2a or alfa-2b + ribavirin.
  Interventions: Biological: Peginterferon alfa-2b; Drug: Ribavirin; Biological: Peginterferon alfa-2a

INTERVENTIONS:
Biological: Peginterferon alfa-2b — Peginterferon alfa-2b administered in accordance with approved labeling
  Other Names: SCH 054031; PegIntron
Drug: Ribavirin — Ribavirin administered in accordance with approved labeling
  Other Names: SCH 018908; Copegus; Rebetol; Virazole; RBV
Biological: Peginterferon alfa-2a — Peginterferon alfa-2a administered in accordance with approved labeling
  Other Names: Pegasys

SUMMARY:
The goal of this study is to elucidate the reasons why patients with chronic hepatitis C (CHC) would not be considered eligible for antiviral treatment. The study is conducted in common clinical practice at approximately 54 sites in Italy. Patients deemed eligible for antiviral therapy will be treated at the discretion of the physician with either peginterferon alfa-2a or peginterferon alfa-2b, both in combination with ribavirin, in accordance with approved labeling. A secondary objective of this study is to define "treatment failure" and to evaluate the reasons for treatment discontinuation.

DETAILED DESCRIPTION:
Probability sampling: Consecutive adult patients with chronic hepatitis C in clinical practice at approximately 54 sites in Italy will be included in the study. The decision as to treatment choice falls at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign an Informed Consent
* Male and female patients >=18 years of age with Chronic Hepatitis C
* Not previously treated with Peg-Interferons
* Positive for serum hepatitis C virus (HCV)-ribonucleic acid (RNA)

Exclusion Criteria:

* Previous treatment with peginterferon
* Participation in a therapeutic Good Clinical Practice (GCP) clinical study within 30 days prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients with chronic hepatitis C seen in common clinical practice at approximately 54 sites in Italy. Treatment for hepatitis C is determined at the local site (pegylated interferon a or b/ribavirin).
Sampling Method: Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

REFERENCES:
- [Derived] Vukotic R, Gamal N, Andreone P. Prospective, observational real-life study on eligibility for and outcomes of antiviral treatment with peginterferon alpha plus ribavirin in chronic hepatitis C. Dig Liver Dis. 2015 Feb;47(2):151-6. doi: 10.1016/j.dld.2014.11.002. Epub 2014 Nov 13. PMID 25483909

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Chronic Hepatitis C (CHC): Peginterferon-naïve participants with chronic hepatitis C (CHC) seen in general clinical practice in Italy.
Period: Overall Study
Arm/Group | Participants With Chronic Hepatitis C (CHC)
Started | 1128
Received Antiviral Treatment | 500
Completed | 326 (Completed defined as participants who completed anti-viral treatment.)
Not Completed | 802
Not completed — Excluded - Prior Use of Peginterferon | 7
Not completed — Excluded - Hepatitis C Virus Negative | 3
Not completed — Not Eligible for Treatment | 431
Not completed — Participant Refused Treatment | 89
Not completed — Never Started Treatment | 89
Not completed — Unknown; No Data Sources Available | 9
Not completed — Physician Decision | 116
Not completed — Withdrawal by Subject | 45
Not completed — Investigator + Participant Decision | 13

BASELINE CHARACTERISTICS:
Groups:
- Participants With Chronic Hepatitis C (CHC): Peginterferon-naïve participants with CHC seen in general clinical practice in Italy.
Arm/Group | Participants With Chronic Hepatitis C (CHC)
Number analyzed (Participants) | 1118
Age, Customized [Number; unit: participants]
  18-29 years | 51
  30-39 years | 119
  40-49 years | 244
  50-59 years | 211
  60-69 years | 263
  70-79 years | 210
  ≥80 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 541
  Male | 577

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Not Eligible for Antiviral Treatment by Reason for Non-eligibility
Description: Investigators recorded their reasons for not prescribing anti-viral treatment. More than one reason leading to non-eligibility could be presented for the same participant.
Time Frame: Measured at baseline
Population: 431 of the 1118 participants were determined to be non-eligible for antiviral therapy by Investigator decision.
Measure: Number; unit: participants
Arm/Group | Participants With Chronic Hepatitis C (CHC)
Number analyzed (Participants) | 431
participants
  Age | 144
  Mild disease | 77
  Substance abuse history | 17
  Treatment postponed | 7
  Genotype | 2
  Comorbidity | 139
  Liver problems | 41
  Problems with previous treatment | 4

2. Secondary Outcome: Number of Participants Discontinued From Treatment by Reason for Discontinuation
Description: Investigators recorded reasons for treatment discontinuation.
Time Frame: 24 weeks after the end of treatment (total of 48 to 72 weeks)
Population: Reasons for treatment discontinuations were recorded by Investigators for 174 of the 500 treated participants.
Measure: Number; unit: participants
Arm/Group | Participants With Chronic Hepatitis C (CHC)
Number analyzed (Participants) | 174
participants
  Disease worsening | 3
  Side effects | 27
  Non response | 44
  Adverse effect | 32
  Administrative reason | 5
  Virological response | 22
  Other reasons | 5

3. Secondary Outcome: Number of Participants With Treatment Failure by Reason for Failure
Description: Investigators recorded reasons for treatment failure whether or not treatment was completed.
Time Frame: 24 to 48 weeks
Population: 132 of the 500 treated participants failed treatment per Investigator assessment.
Measure: Number; unit: participants
Arm/Group | Participants With Chronic Hepatitis C (CHC)
Number analyzed (Participants) | 132
participants
  Disease relapse | 71
  Non-responder | 61

ADVERSE EVENTS:
Description: 500 participants on this study were treated with either PegInterferon alfa-2a or alfa-2b/+ ribavirin per facility guidelines but treatment drugs were not recorded for this study. Adverse events (AEs) were collected for participants treated with any Sponsor product, but not with other company products; therefore, the AEs are disclosed at 0% level.
Arm/Group | Participants With Chronic Hepatitis C (CHC)
Serious Adverse Events (participants affected / at risk) | 6/500
Other Adverse Events (participants affected / at risk) | 169/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Chronic Hepatitis C (CHC) (N=500)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Chronic Hepatitis C (CHC) (N=500)
Anaemia (Blood and lymphatic system disorders) | 64 (65)
Haemoglobinaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 10 (10)
Neutropenia (Blood and lymphatic system disorders) | 23 (23)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)
Tachycardia (Cardiac disorders) | 3 (3)
Deafness (Ear and labyrinth disorders) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 4 (4)
Hypothyroidism (Endocrine disorders) | 7 (7)
Chalazion (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7)
Aerophagia (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 47 (47)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Hyperpyrexia (General disorders) | 7 (7)
Influenza like illness (General disorders) | 19 (19)
Injection site reaction (General disorders) | 2 (2)
Irritability (General disorders) | 3 (3)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 19 (19)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Tooth abscess (Infections and infestations) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Serum ferritin increased (Investigations) | 1 (1)
Thyroid function test abnormal (Investigations) | 1 (1)
Weight decreased (Investigations) | 12 (12)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Insulin resistance (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 12 (12)
Paraesthesia (Nervous system disorders) | 2 (2)
Polyneuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 11 (11)
Apathy (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 8 (8)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 11 (11)
Mood altered (Psychiatric disorders) | 1 (1)
Nervousness (Psychiatric disorders) | 3 (3)
Panic attack (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspoenia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 14 (14)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Trichorrhexis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator agrees not to publish or publicly present any interim results of the Study without prior written consent of the sponsor. The principal investigator further agrees to provide 45 days written notice to the sponsor prior to submission for publication or presentation to permit the sponsor to review copies of abstracts or manuscripts for publication.